CLINICAL TRIAL: NCT06515886
Title: Characterizing the Inflammation Around Dental Implants: Bacterial Infection, Hypersensitivity or Both?
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Nicholas Makhoul, Associate professor and Associate Dean of Post-Graduate Dental Education, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 20227639
Record Dates: First submitted 2024-07-15; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Dental Implant Failed; Implant Complication; Implant Site Infection; Implant Site Reaction
Keywords: Dental implant; Peri-implant inflammation; Inflammatory mediators; Bacterial infection; Hypersensitivity; peri-implantitis
MeSH Terms: conditions — Bacterial Infections; Hypersensitivity; Peri-Implantitis | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Peri-implant crevicular fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dental implants: Intra-oral photograph
  Sample of Peri-implant Crevicular fluid
  Clinical Examination
  Peri-apical x-ray
  Interventions: Diagnostic Test: Clinical Examination; Procedure: Peri-implant crevicular fluid

INTERVENTIONS:
Diagnostic Test: Clinical Examination — Clinical examination of a dental implant
Procedure: Peri-implant crevicular fluid — Collection of a sample of peri-implant crevicular fluid

SUMMARY:
The use of titanium dental implants has become a common modern treatment to restore teeth. Although the success rate of dental implants is high, inflammation around the dental implant still occurs. The current study will investigate if the inflammation around the implant is due to bacterial infection, hypersensitivity or both.

DETAILED DESCRIPTION:
The objective of the study is to:

1. Establish the levels of cytokines in peri-implant crevicular fluid and test the levels of cytokines associated with hypersensitivity (Type 2: Interleukin-4 [IL-4], Interleukin-5 [IL-5], and Interleukin-13 [IL-13]) and bacterial infection (Type 1 and 3: Interleukin-1 alpha [IL-1α], Interleukin-2 [IL-2], Interleukin-6 [IL-6], Interleukin-8 [IL-8], Interleukin-10 [IL-10], Interleukin-12 [IL-12], Interleukin-17 [IL-17], Granulocyte-Macrophage Colony-Stimulating Factor [GM-CSF], Interferon-gamma [IFN-γ], Tumor Necrosis Factor-alpha [TNF-α]) between healthy implants and inflamed implants (mucositis and peri-implantitis).
2. Compare the levels of Matrix Metalloproteinases (MMPs: MMP-1, MMP-2, and MMP-9) and Receptor Activator of Nuclear Factor Kappa-Β Ligand (RANKL) associated with tissue destruction and bone loss between healthy and inflamed implants.

ELIGIBILITY:
Inclusion Criteria:

* Received at least one functional implant (implant restored with a prothesis);
* Did not receive peri-implant mucositis and peri-implantitis treatment in the past three months.

Exclusion criteria:

* Dental records with incomplete information;
* Individuals with a weak immune system or chronic disease such as diabetes, heart, lung or kidney disease;
* Pregnant women;
* Individuals undergoing orthodontic therapy and those who have oral piercing.
* History of diseases that modify or suppress the immune and inflammatory response, including rheumatoid arthritis, diabetes, lupus, and inflammatory bowel disease and metastatic cancer;
* Taking medications that cause antiresorptive osteonecrosis of the jaw (including any dose of intravenous bisphosphonates, oral bisphosphonate intake for more than three years, receptor activator of nuclear factor kappa-B ligand inhibitors, or antiangiogenic medications);
* Taking medications known to induce gingival hyperplasia including anticonvulsants, immunosuppressants, or calcium channel blockers;
* Taking steroid medications, systemic or local antibiotics in the last three months (as this may affect the interleukins activity);
* Received radiation therapy to the head and neck or chemotherapy;
* Received treatment to manage an inflamed implant, including management of peri-implantitis and peri-implant mucositis in the last three months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This cross-sectional study is carried out at McGill University Health Center (MUHC)-Montreal General Hospital Oral and Maxillofacial Clinic. The electronic dental records database at the MUHC Montreal General Hospital Oral and Maxillofacial Clinic is screened to identify potentially eligible participants. Individuals who had a functional implant (implant restored with a prosthesis) placed between 2010 and 2022 were reviewed. Eligible individuals are contacted and invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Levels of cytokines in peri-implant crevicular fluid associated with hypersensitivity | September 2022 - December 2024
  Measure the levels of IL-4, IL-5, and IL-13 in the peri-implant crevicular fluid to assess hypersensitivity responses between healthy implants and inflamed implants (mucositis and peri-implantitis).
  The measured unit is pg/ml.
Levels of cytokines in peri-implant crevicular fluid associated with bacterial infection | September 2022 - December 2024
  Measure the levels of IL-1α, IL-2, IL-6, IL-8, IL-10, IL-12, IL-17, TNF-α, GM-CSF, and IFN-γ in the peri-implant crevicular fluid to assess bacterial responses between healthy implants and inflamed implants (mucositis and peri-implantitis).
  The measured unit is pg/ml.
Levels of Matrix Metalloproteinases in peri-implant crevicular fluid | September 2022 - December 2024
  Measure the levels of MMP-1, MMP-2, and MMP-9 in the peri-implant crevicular fluid to assess hypersensitivity responses between healthy implants and inflamed implants (mucositis and peri-implantitis).
  The measured unit is pg/ml.
Levels of RANKL in peri-implant crevicular fluid | September 2022 - December 2024
  Measure the levels of RANKL in the peri-implant crevicular fluid to assess hypersensitivity responses between healthy implants and inflamed implants (mucositis and peri-implantitis).
  The measured unit is pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Allah Madi Dr, Principal Investigator — McGill University; Nicholas Makhoul Dr, Study Director — McGill University; Jocelyne Feine Dr, Study Director — McGill University
Locations (1):
- Montreal General Hospital - Oral & Maxillofacial Surgery Clinic, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided